CLINICAL TRIAL: NCT01474941
Title: A Phase 1, Randomized, Double-Blind, Parallel, Placebo-Controlled, Multiple-Dose Escalation Study To Investigate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of A Modified-Release Formulation Of PF-04620110 In Otherwise Healthy Overweight Or Obese Adult Subjects
Brief Title: A Study Of PF-04620110 As A Modified-Release Formulation In Healthy Overweight Or Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: B0961011
Record Dates: First submitted 2011-06-09; First posted 2011-11-18 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: Multiple Dose Study Overweight Healthy Subjects Body Weight Modified-Release Formulation
MeSH Terms: interventions — PF-04620110

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 5 mg QD PF-04620110 or Placebo (Experimental)
  Interventions: Drug: PF-04620110 or Placebo
- 5 mg BID PF-04620110 or Placebo (Experimental)
  Interventions: Drug: PF-04620110 or Placebo
- Optional Arm, PF-04620110 or Placebo (Experimental)
  Interventions: Drug: PF-04620110 or Placebo

INTERVENTIONS:
Drug: PF-04620110 or Placebo — Multiple oral doses of 5 mg PF-04620110 as a modified-release formulation or placebo once daily for 2 weeks
  Arms: 5 mg QD PF-04620110 or Placebo
Drug: PF-04620110 or Placebo — Multiple oral doses of 5 mg PF-04620110 as a modified-release formulation or placebo twice daily for 2 weeks
  Arms: 5 mg BID PF-04620110 or Placebo
Drug: PF-04620110 or Placebo — Repeat Arm 1 or Arm 2
  Arms: Optional Arm, PF-04620110 or Placebo

SUMMARY:
The primary purpose of this trial is to evaluate the safety and tolerability, pharmacokinetics and pharmacodynamics, of multiple oral doses of PF-04620110 as a modified-release formulation.

DETAILED DESCRIPTION:
To evaluate the safety and tolerability, pharmacokinetics (PK), and pharmacodynamics, of multiple oral doses of PF-04620110 as a modified-release formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 27 to 35 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease or clinical findings at screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2011-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability data: number of subjects with adverse events and Laboratory Test Values of Potential Clinical Importance, Changes fro baseline in pulse rate, blood pressure and ECG measurements over 14 days. | 2 weeks
Profile of Pharmacokinetics: timeframe 0, 0.5, 1,2.5, 4.5, 6.5, 8.5, 10, 10.5, 11, 12.5, 14.5, 16.5 and 24 hr on Days 1 and 14. 24, 48, 72, 96, 120, 144 and 216 hrs post first dosing | 2 weeks
PK parameters: Area under the Concentration-Time Curve (AUC), Maximum Observed Plasma Concentration (Cmax), Time to Reach Maximum Observed Plasma Concentration (Tmax), Apparent Oral Clearance (CL/F), Accumulation Ratios (Cmax,ss/Cmin,ss, AUC | 2 weeks
(0-24,ss)/AUC(0-24,sd) andCmax,ss/Cmax,sd) | 2 weeks
Glucose response: 24-hour (AUC(0-24)/24), post-MMTT (AUC(0.5-4.5)/4), post-lunch (AUC(4.5-10.5)/6) and post-dinner (AUC(10.5-16.5)/6) weighted mean average glucose on Days 0 and 14; fasting plasma glucose | 2 weeks
Insulin response: 24-hour (AUC(0-24)/24), post-MMTT (AUC(0.5-4.5)/4), post-lunch (AUC(4.5-10.5)/6) and post-dinner (AUC(10.5-16.5)/6) weighted mean average insulin on Days 0 and 14; fasting plasma insulin | 2 weeks
total GLP-1 response: 24-hour (AUC(0-24)/24), post-MMTT (AUC(0.5-4.5)/4), post-lunch (AUC(4.5-10.5)/6) and post-dinner (AUC(10.5-16.5)/6) weighted mean average total GLP-1 on Days 0 and 14; fasting total GLP-1 | 2 weeks
net triglycerides response: 24-hour (AUC(0-24)/24), post-MMTT (AUC(0.5-4.5)/4), post-lunch (AUC(4.5-10.5)/6) and post-dinner (AUC(10.5-16.5)/6) weighted mean average net triglycerides on Days 0 and 14; fasting plasma net triglycerides | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0961011&StudyName=A%20Study%20Of%20PF-04620110%20As%20A%20Modified-Release%20Formulation%20In%20Healthy%20Overweight%20Or%20Obese%20Subjects%20%20